CLINICAL TRIAL: NCT01946633
Title: Remote-controlled Capsule Endoscopy: a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xinying wang, Associate Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GNF-NaviCam-001
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Ulcer; Gastric Polyp
MeSH Terms: conditions — Stomach Ulcer; Polyposis, Gastric

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esophagogastroduodenoscopy（ECG） (Experimental): n=15
  Interventions: Device: magnetic-controlled capsule endoscopy(Navicam)

INTERVENTIONS:
Device: magnetic-controlled capsule endoscopy(Navicam)

SUMMARY:
The present study is a feasibility study to assess the safety and efficacy of wireless capsule endoscope and compare the data obtained with those obtained by using a conventional esophagogastroduodenoscopy.

The product was developed and manufacture in China.(the NaviCam. AKC-1.China)

ELIGIBILITY:
Inclusion Criteria:

* upper abdominal symptoms (≥1 year )
* surveillance gastroscopy for known gastric ulcer or polyps
* history of gastric ulcer or polyps （≤1w）at Nanfang Hospital were enrolled.

Exclusion Criteria:

* dysphagia
* suspected or documented digestive tract malformation ,obstruction, strictures or fistula
* acute upper GI bleeding, acute enteritis, acute ischemia disease
* history of abdominal operations
* impaired renal function, congestive heart failure
* patients with critical condition or mental illness
* patients with, known allergy to polymer material or antifoam agent
* patients with cardiac pacemakers or other implanted electromedical devices，magnetic resonance imaging ( mri) examination in 7 days
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
the percentage of complete visualization of anatomic landmarks | 2 year
  the percentage of patients in whom there was complete visualization of the gastric surface in the antrum, body, and fundus and identification of the cardia and pylorus
examination time and the percentage of abnormal finding | 2 year
  examination time and the percentage of abnormal findings seen on gastroscopy that were reproducible by capsule endoscopy

SECONDARY OUTCOMES:
adverse effect | 2 year
  any discomfort like chest pain, nausea will be documented. capsule retention（defined as not extrusion in 14 days）will be documented.
Acceptability | 2 year
  Acceptability to patients was assessed by means of a questionnaire, with ratings on a scale of 0 to 10 and examination chosen for next time. completed in the recovery room immediately after capsule examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Gastroenterology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Keller J, Fibbe C, Volke F, Gerber J, Mosse AC, Reimann-Zawadzki M, Rabinovitz E, Layer P, Schmitt D, Andresen V, Rosien U, Swain P. Inspection of the human stomach using remote-controlled capsule endoscopy: a feasibility study in healthy volunteers (with videos). Gastrointest Endosc. 2011 Jan;73(1):22-8. doi: 10.1016/j.gie.2010.08.053. Epub 2010 Nov 9. PMID 21067740
- See also: Inspection of the human stomach using remote-controlled capsule endoscopy: a feasibility study in healthy volunteers — http://www.ncbi.nlm.nih.gov/pubmed/21067740